CLINICAL TRIAL: NCT04884724
Title: Effects of Adaptive Dance Exercise Program on Trunk Control, Balance and Functional Mobility in Children and Adolescents with Cerebral Palsy
Brief Title: Adaptive Dance Exercise Program on Trunk Control, Balance and Functional Mobility in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Asena Yekdaneh, University Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAGulnergiz
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Trunk Control; Mobility; Adaptive Dance; Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adaptive Dance Exercise Group (Experimental): In addition to the routine physiotherapy programs received in the rehabilitation center for children and adolescents with cerebral palsy, an adaptive dance exercise program will be applied 2 days a week in the rehabilitation center for 5 weeks and online for 3 weeks in the presence of a physiotherapist. The duration of each session of the adaptive dance exercises to be applied is planned to be 45-60 minutes. It is planned that the adaptive dance exercises to be applied will be accompanied by the selected song.
  Before and after the 8-week exercise program, the participants' trunk stabilization, balance, functional mobility and quality of life will be questioned with determined questionnaires and tests.
  Interventions: Other: Adaptive Dance Exercise Program
- Control Group (No Intervention): Children and adolescents diagnosed with Cerebral Palsy will continue their routine physiotherapy and rehabilitation programs in the rehabilitation center. At the beginning of the study and after 8 weeks, the participants' trunk stabilization, balance, functional mobility and quality of life will be questioned with determined questionnaires and tests.

INTERVENTIONS:
Other: Adaptive Dance Exercise Program — It is planned to include balance, stabilization, mobility, speed and rhythm activities for the exercises applied in Cerebral Palsy rehabilitation and based on the principles of motor learning, and to apply the dance steps and figures to be applied with visual and auditory stimuli.
  Arms: Adaptive Dance Exercise Group

SUMMARY:
The human body needs a system to control and coordinate its action plan in order to perform an effective action. This system works irregularly or inappropriately in people with Cerebral Palsy (CP). An alternative to controlling these disorders is automatic movement modulation such as dance. Dance, whose main purpose is to achieve a satisfying motor performance, increases motor learning with sensory, perceptual and emotional components. Although the effects of dance therapy on functionality, balance and participation in people with CP have been previously examined in the literature, it has been reported that the evidence is insufficient and more studies are needed. The aim of this study is to examine the effects of adaptive dance exercise program on trunk control, balance and functional mobility in children and adolescents with Cerebral Palsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cerebral Palsy
* Volunteer
* Ages between of 6-18 years
* Gross Motor Function Classification System (GMFCS) Level 1 and Level 2
* To have cognitive skills to understand and apply adaptive dance exercises to be given.

Exclusion Criteria:

* Participants diagnosed with Cerebral Palsy having cognitive disorders
* Participants diagnosed with Cerebral Palsy having vision or hearing problems
* Participants diagnosed with Cerebral Palsy have a history of trauma such as botox or muscle relaxation operation and / or fracture at least 6 months before participating in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS). Change is being assessed. | Change from Baseline TCMS Score at 8 weeks
  TCMS consists of static sitting balance, dynamic sitting control (Selective motor control and dynamic reaching) sections. The scale consists of 15 items in total and is divided into five, seven and three items. All items are evaluated bilaterally and scored on a 2, 3 or 4 point rank scale. TCMS total score is between 0-58 and the higher the score, the better the performance. Participants' trunk stabilization will be evaluated with TCMS.
Pediatric Balance Scale (PBS). Change is being assessed. | Change from Baseline PBS Score at 8 weeks
  The five-level consists of 14 elements such as sitting balance, standing balance, standing up from sitting, moving from standing to sitting, transfers, stepping, reaching, turning and jumping. Each item is scored between 0-4 points. High scores indicate better performance. Participants' balance will be evaluated with PBS.
Time Up and Go (TUG). Change is being assessed. | Change from Baseline TUG Score at 8 weeks
  The participant sitting on the floor without arm support, hip and knee flexed at 90 degrees and feet on the ground are asked to stand up, walk 3 meters, turn around and sit on the chair. The test is applied 3 times, the time is recorded and the average of 3 trials is taken. Participants' functional mobility will be evaluated with TUG.

SECONDARY OUTCOMES:
Pediatric Outcomes Data Collection Instrument (PODCI). Change is being assessed. | Change from Baseline PODCI Score at 8 weeks
  PODCI has 2 parent forms (child and adolescent) and adolescent forms consisting of the same questions. The test is a Likert-type scale and consists of 5 parts: Upper Extremity Functions-UEF, Physical Function and Sport-FFS, Transfer and Basic Mobility-TM, Pain-RA and Happiness / Satisfaction-MM, as well as Expectations-TB section where expectations from treatment are questioned. Each section is calculated between 0-100. Participants' quality of life will be evaluated with PODCI.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Asena Yekdaneh, Pt.,MSc., Principal Investigator — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Istanbul
  - Işıl Özel Eğitim ve Rehabilitasyon Merkezi, Istanbul

IPD SHARING:
Plan to Share IPD: No